CLINICAL TRIAL: NCT03883945
Title: A Randomized, Double-Blind, Vehicle-Controlled, Parallel-Group, Dose-Escalation Study to Evaluate the Safety and Pharmacokinetics of Intradermally Administered AIV001 in Subjects With Papulopustular Rosacea
Brief Title: A Safety and Efficacy Study to Evaluate Rosacea
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Sponsor deprioritization
Sponsor: AiViva BioPharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AIV001-R01
Record Dates: First submitted 2019-03-16; First posted 2019-03-21 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Papulopustular Rosacea
Keywords: rosacea
MeSH Terms: conditions — Rosacea

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, vehicle-controlled, parallel-group, dose-escalation study evaluating study medication versus vehicle in each of 4 sequentially enrolled cohorts
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Study medication will be administered by the Treating Investigator. Safety and efficacy measures will be evaluated by the masked Evaluating Investigator.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (8):
- Cohort 1 - vehicle (Placebo Comparator): Subjects randomized to vehicle will receive vehicle administration to the target area.
  Interventions: Drug: Vehicle
- Cohort 1 - 0.033% (Active Comparator): Subjects randomized to vehicle will receive AIV001 0.033% administration to the target area.
  Interventions: Drug: AIV001
- Cohort 2 - vehicle (Placebo Comparator): Subjects randomized to vehicle will receive vehicle administration to the target area.
  Interventions: Drug: Vehicle
- Cohort 2 - 0.1% (Active Comparator): Subjects randomized to vehicle will receive AIV001 0.01% administration to the target area.
  Interventions: Drug: AIV001
- Cohort 3 - vehicle (Placebo Comparator): Subjects randomized to vehicle will receive vehicle administration to the target area.
  Interventions: Drug: Vehicle
- Cohort 3 - 0.3% (Active Comparator): Subjects randomized to vehicle will receive AIV001 0.03% administration to the target area.
  Interventions: Drug: AIV001
- Cohort 4 - vehicle (Placebo Comparator): Subjects randomized to vehicle will receive vehicle administration to the target area.
  Interventions: Drug: Vehicle
- Cohort 4 - 1% (Active Comparator): Subjects randomized to vehicle will receive AIV001 0.03% administration to the target area.
  Interventions: Drug: AIV001

INTERVENTIONS:
Drug: AIV001 — intradermal injection
  Arms: Cohort 1 - 0.033%; Cohort 2 - 0.1%; Cohort 3 - 0.3%; Cohort 4 - 1%
Drug: Vehicle — intradermal injection
  Arms: Cohort 1 - vehicle; Cohort 2 - vehicle; Cohort 3 - vehicle; Cohort 4 - vehicle

SUMMARY:
To evaluate the safety, efficacy, and pharmacokinetic profile of ascending concentrations of the study medication compared with vehicle in subjects with rosacea.

DETAILED DESCRIPTION:
This is primarily a safety study to evaluate the safety of AIV001 when administered to subjects with rosacea. Exploratory efficacy measures will also be collected as well as pharmacokinetic profiles.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 18 and 65 year with rosacea, 10 to 30 papules and pustules (at least 5 lesions within the treatment area on each facial side), and < 2 nodules
* Presence of moderate to severe persistent erythema
* Total body weight >45 kg

Exclusion Criteria:

* Presence of any skin condition on the face that would interfere with the diagnosis or assessment of rosacea
* Extremely dark skin type that would confound the digital analysis of erythema (eg, Fitzpatrick Skin Type 5 or 6)
* Excessive facial hair (eg, beards, sideburns, moustaches, etc.), birthmarks, or tattoos that would interfere with diagnosis or assessment of rosacea
* Use of tobacco- or nicotine-containing products in excess of the equivalent of 5 cigarettes per day.
* Pregnant or nursing females; females of childbearing potential who are unwilling or unable to use an acceptable method of non-hormonal contraception as outlined in this protocol from at least 14 days prior to start of treatment.
* Hypersensitivity or allergy to axitinib or any other component of the study treatment
* Use within 6 months prior to baseline and during the study of oral retinoids (eg, Accutane®) or therapeutic vitamin A supplements of greater than 10,000 units/day (multivitamins are allowed).
* Use within 6 weeks prior to baseline and during the study of vasodilators or α-adrenergic receptor-blocking agents.
* Use within 1 month prior to baseline and during the study of 1) topical retinoids to the face, 2) systemic antibiotics know to have an impact on the severity of facial rosacea (eg, containing tetracycline and its derivatives, erythromycin and its derivatives, sulfamethoxazole, or trimethoprim), 3) systemic corticosteroids, or 4) facial light-based therapies

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-07 (Estimated); Primary Completion 2022-07 (Estimated); Study Completion 2022-08 (Estimated)

PRIMARY OUTCOMES:
Rate of Adverse Events | Day 1 through Day 84
  The occurrence of adverse events will be collected and reported using MedDRA to code. Description, start and end dates, and severity will be recorded.

SECONDARY OUTCOMES:
Efficacy evaluated by the Investigator using the Investigator Global Assessment Scale | Day 1 through Day 84
  Evaluation of rosacea within the treatment area. 0 = clear (No papules and/or pustules; no or residual erythema; no or mild to moderate telangiectasia), 1 = minimal (Rare papules and/or pustules; residual to mild erythema; mild to moderate telangiectasia), 2 = mild (Few papules and/or pustules; mild erythema; mild to moderate telangiectasia), 3 = mild to moderate (Distinct number of papules and/or pustules; mild to moderate erythema; mild to moderate telangiectasia), 4 = moderate (Pronounced number of papules and/or pustules; moderate erythema; mild to moderate telangiectasia), 5 = moderate to severe (Many papules and/or pustules; occasionally with large inflamed lesions; moderate erythema; moderate degree of telangiectasia), and 6 = severe (Numerous papules and/or pustules, occasionally with confluent areas of inflamed lesions; moderate or severe erythema; moderate or severe telangiectasia). Scores of 0 or 1 are considered success.
Efficacy evaluated by the Investigator by performing Inflammatory Lesion Counts | Day 1 through 84
  The number of inflammatory lesions is a static measure of the number of papules or pustules present within the treatment area.
Evaluation of Erythema and Topography using Standardized Photography | Day 1 through 84
  Photographs using standardized equipment will be taken and uploaded onto the vendor's server. The vendor will then use proprietary software to measure the amount of redness and the topography of the lesions within the treatment area.

CONTACTS AND LOCATIONS:
Overall Officials: Mitchell Goldman, MD, Principal Investigator — West Dermatology
Locations (1):
- Cosmetic Laser Dermatology, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No